CLINICAL TRIAL: NCT00096564
Title: Functional MRI Study of Brain Activation With Observation of Facial Expressions
Brief Title: Brain Activities Associated With Different Facial Expressions Using Blood Oxygenation Level Dependent Functional MRI
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050032; 05-N-0032
Record Dates: First submitted 2004-11-10; First posted 2004-11-11 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-08-20

CONDITIONS: Healthy
Keywords: Mirror Neuron; Urge; Statistical Parametric Mapping; Healthy Volunteer; HV

SUMMARY:
Objectives: The purpose of this study is to identify areas of brain activation during the urge to yawn. Little is known about how yawning is suppressed, or why yawning often occurs in response to seeing another person yawn (contagious yawning). Contagious yawning is similar to other contagious motor programs, such as the greater urge Tourette subjects feel to tic when seeing repetitive movements or other subjects' tics, the urge to scratch when discussing itching and scratching, or the urge to urinate when hearing running water. Hypothetically, the urge or the suppression of this urge is modulated by a common cortical circuit implicated in Tourette syndrome. We plan to use functional magnetic resonance imaging (fMRI) to identify the pattern of blood oxygenation level-dependent (BOLD) activation in the brain when normal volunteers feel the urge to yawn.

Study Population: We intend to study 25 normal, right-handed, healthy volunteers.

Study Design: Using an event-related design, we will scan subjects, using the same 3T fMRI scanner, while showing a video of a person yawning, gaping, coughing, or doing nothing. Each of these four action stimuli will last for four seconds, with varying interstimulus intervals. Each video set will contain all actions displayed ten times pseudorandomly. Two data sets will be collected from each subject and will be separated by a brief rest period. Subjects will be instructed before the scan to watch a videotaped person perform various behaviors, without detailing the specific actions. So as not to influence their natural response to the yawning stimulus, we will instruct them only to keep their head still. The variable of interest will be the activation during urge-generation, contrasted with other control stimuli. A survey will be administered for informational purposes following the scan to assess the subjects' general impression of their susceptibility to yawning, whether they yawned in the scanner, whether they suppressed the urge to yawn, and if the urge to yawn increased or decreased with the repetition of the yawning segment.

Outcome Measures: The primary outcome of this study is the activation of brain structures in response to viewing another person yawning. In particular, we are interested in the activation of the anterior cingulate cortex, parietal operculum, insula, supplementary motor area, and dorsolateral prefrontal cortex as these are areas implicated in the urge to move in response to either internal (as in Tourette syndrome) or external (as in itching from histamine injection) states. Since the urge to yawn is the process of interest, suppression of yawning is not relevant to the fMRI analysis.

DETAILED DESCRIPTION:
Purpose of this study

This study will look at how perception and observation of various facial expressions may affect the way different areas of the brain function. We hope to gain a greater understanding of abnormal movements, such as tics, by investigating how facial expressions affect the brain.

Background Information

This study is based on prior research that focuses on the activity and changes in different areas of the brain depending on what people see others around them doing. An example is the feeling of empathy one might have when looking at a sad face, or anxiety and fear when looking at an angry face.

Who is the Study Population?

20 healthy, right-handed men and women

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects age 18 and older.

Subjects willing to abstain from caffeine or alcohol for 48 hours prior to the fMRI scanning.

EXCLUSION CRITERIA:

Subjects with any abnormal findings on neurological exam.

Subjects with a positive urine pregnancy test.

Subjects who are pregnant.

Subjects with any finding on the MRI safety questionnaire which prevents them from safely undergoing an MRI scan.

Subjects with any history of brain tumor, stroke, head trauma or a vascular malformation as obtained by history or from imaging studies.

Subjects with any history of a severe medical condition, such as cardiovascular disease, which would prevent them from lying flat for up to 60 minutes.

Subjects without the capacity to give informed consent.

Subjects with claustrophobia or other restrictions which prevent them from undergoing a scan in a confined space for up to 60 minutes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2004-11-09; Study Completion 2008-08-20

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Argiolas A, Melis MR. The neuropharmacology of yawning. Eur J Pharmacol. 1998 Feb 5;343(1):1-16. doi: 10.1016/s0014-2999(97)01538-0. PMID 9551709
- [Background] Askenasy JJ. Is yawning an arousal defense reflex? J Psychol. 1989 Nov;123(6):609-21. doi: 10.1080/00223980.1989.10543014. PMID 2558182
- [Background] Athwal BS, Berkley KJ, Hussain I, Brennan A, Craggs M, Sakakibara R, Frackowiak RS, Fowler CJ. Brain responses to changes in bladder volume and urge to void in healthy men. Brain. 2001 Feb;124(Pt 2):369-77. doi: 10.1093/brain/124.2.369. PMID 11157564